CLINICAL TRIAL: NCT00363922
Title: Rehabilitation After Coronary Bypass Grafting: Home Based Rehabilitation Versus Rehabilitation in Institution and Rehabilitation in Institution Versus Out-patient Rehabilitation at the Hospital
Brief Title: Rehabilitation After Coronary Bypass Grafting. Comparison of Different Types of Rehabilitation Programs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2006.2070
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass [E04.100.376.719.332]
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rehabilitation; Academies and Institutes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rehabilitation in institution
  Interventions: Behavioral: Rehabilitation in institution
- 2 (Active Comparator): Rehabilitation at home
  Interventions: Behavioral: Rehabilitation at home; Behavioral: Out-patient rehabilitation at the hospital

INTERVENTIONS:
Behavioral: Rehabilitation in institution — Rehabilitation in institution for four weeks. Subjects follow standard rehabilitation in the center.
  Arms: 1
Behavioral: Rehabilitation at home — Subjects get a written prescription of exercise training, diet, etc. to follow at home.
  Arms: 2
Behavioral: Out-patient rehabilitation at the hospital — This intervention was removed. We never got time to randomize subjects into this category. We had planned to randomize patients from one hospital to either Rehabilitation in institution (rehab center) or rehabilitation at the hospital (out patient). And also patients from another hospital to either rehabilitation in institution (rehab centre) or rehabilitation at home. We have only managed to start the study in this second hospital so far (due to maternity leave and limited time to finish a PhD)
  Arms: 2

SUMMARY:
The purpose of this study is to compare different types of rehabilitation after coronary bypass surgery. The investigators wish to compare rehabilitation in an institution for four weeks with a home based rehabilitation. They also wish to compare rehabilitation in an institution for four weeks with a rehabilitation program were the patients live at home but visit the hospital twice a week for twelve week. The investigators will measure the patients' physical capacity by measuring their maximal oxygen consumption. The investigators will also analyze their blood and their endothelian function (how well their arteries dilate).

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass

Exclusion Criteria:

* Significant lung disease
* Drug abuse
* Pregnancy
* Major physical impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | At baseline and after 6 months

SECONDARY OUTCOMES:
Blood analyses (different markers for cardiovascular risk and endothelian function) | At baseline and after 6 months
Endothelian function (flow mediated dilatation) | At baseline and after 6 months
Quality of life (SF36 and MacNew) | At baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Trine T. Moholdt, cand.polit, Principal Investigator — National Taiwan Normal University
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Moholdt T, Bekken Vold M, Grimsmo J, Slordahl SA, Wisloff U. Home-based aerobic interval training improves peak oxygen uptake equal to residential cardiac rehabilitation: a randomized, controlled trial. PLoS One. 2012;7(7):e41199. doi: 10.1371/journal.pone.0041199. Epub 2012 Jul 18. PMID 22815970